CLINICAL TRIAL: NCT02925806
Title: Drug Utilization Study of Trends in Prescriptions for Class REMS ER/LA Opioids and Comparator Products; Evaluation of Drug Utilization Patterns
Brief Title: Evaluation of Drug Utilization Patterns for Extended Release/Long Acting Opioids and Comparator Products
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: ER/LA Opioid REMS Program Companies (RPC) (Industry)
Responsible Party: Sponsor
Other Study IDs: Assessment 6
Record Dates: First submitted 2016-09-28; First posted 2016-10-06 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Opioid Related Disorders; Opiate Addiction; Narcotic Abuse; Drug Abuse
MeSH Terms: conditions — Opioid-Related Disorders; Narcotic-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (4):
- ER/LA opioids included in the class REMS
  Interventions: Other: Non-interventional study - retrospective database review
- IR Opioids
  Interventions: Other: Non-interventional study - retrospective database review
- Celecoxib
  Interventions: Other: Non-interventional study - retrospective database review
- Benzodiazepines
  Interventions: Other: Non-interventional study - retrospective database review

INTERVENTIONS:
Other: Non-interventional study - retrospective database review

SUMMARY:
A drug utilization study will be performed to describe trends in the number of prescriptions and patients for class REMS ER/LA opioids and comparator products.

DETAILED DESCRIPTION:
A drug utilization study will be performed to describe trends in the number of prescriptions and patients for class REMS ER/LA opioids and comparator products.

The specific objectives of the Drug Utilization Study are:

1. To estimate trends by month in the number of prescriptions for a one-year period before, and each month after, the implementation of the REMS
2. To compare average number of prescriptions per 3 month (quarter) period in the 2 years before as compared to the same measure during Implementation and the Active Period
3. To evaluate change by patient characteristics (age group, gender, pay type, prescriber specialty)
4. To compare the trends in prescribing, both number of prescriptions and patients, by prescriber specialty

   These trends and changes over time will be estimated for the following groups of opioids:
   * ER/LA opioids included in the class REMS
   * Comparator products/classes

     * Immediate release (IR) opioids
     * Celecoxib
     * Benzodiazepines
5. To show switches (absolute and rates of switching) from ER/LA opioids to comparator analgesics (IR opioids or celecoxib) with introduction of REMS

ELIGIBILITY:
Inclusion Criteria:

* Subjects filling a prescription for a product of interest during the specified time period will be included.

Exclusion Criteria:

* None

Max Age: 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Subjects filling a prescription for a product of interest as gathered from the IMS National prescription Audit™ and IMS Health, LifeLink™
Sampling Method: Non-Probability Sample
Enrollment: 5575834 (Estimated)
Dates: Primary Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Number of opioid prescriptions filled | Monthly over 54 months
Compare average number of prescriptions per time period in the 2 years before as compared to the same measure in implementation and active periods | Pre REMS Implementation (July 10-June 12)
Compare trends in prescribing, both number of prescriptions and patients, by prescriber specialty | Pre REMS Implementation (July 10-June 12)
Number and Rate of Switches from ER/ LA opioids to comparator analgesics with introduction of REMS | Monthly over 54 months
Compare average number of prescriptions per time period in the 2 years before as compared to the same measure in implementation and active periods | Implementation (July 12-June 13)
Compare average number of prescriptions per time period in the 2 years before as compared to the same measure in implementation and active periods | Active Period (July 13-Dec 14)
Compare trends in prescribing, both number of prescriptions and patients, by prescriber specialty | Implementation (July 12-June 13)
Compare trends in prescribing, both number of prescriptions and patients, by prescriber specialty | Active Period (July 13-Dec 14)